CLINICAL TRIAL: NCT01808937
Title: Immunologic and Genetic Profiles in Subsets of Morphea Patients
Brief Title: Morphea in Adults and Children (MAC) Cohort Study: A Morphea Registry and DNA Repository
Acronym: MAC
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Heidi Jacobe, PROFESSOR, University of Texas Southwestern Medical Center
Other Study IDs: 032007021; STU 112010-028
Record Dates: First submitted 2013-02-25; First posted 2013-03-11 (Estimated); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Scleroderma, Localized; Morphea; Frontal Linear Scleroderma en Coup de Sabre; Scleroderma, Circumscribed; Scleroderma, Linear
MeSH Terms: conditions — Scleroderma, Localized

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Biospecimen Retention: Samples With DNA — serum, WBC, tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Morphea: Those having the condition morphea or other synonymous diagnosis (such as localized scleroderma, linear scleroderma, Parry-Romberg syndrome, en coup de sabre)
  Interventions: Other: Morphea

INTERVENTIONS:
Other: Morphea
  Other Names: Scleroderma, Localized; Scleroderma, Circumscribed; Scleroderma, Linear; Frontal Linear Scleroderma en Coup de Sabre

SUMMARY:
The Morphea in Adults and Children (MAC) cohort is the first registry for both children and adults with morphea (also known as localized scleroderma) in the country. The purpose of the registry is to learn more about morphea, specifically:

* How morphea behaves over time
* How frequently specific problems occur along with morphea (for example, arthritis)
* Whether morphea has an autoimmune background

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have a clinical diagnosis of morphea confirmed by the primary investigator and by histopathological examination.
2. Ages 0-90 years old
3. Children must weigh more than 20 lbs. in order to satisfy Children's Medical Center policy for the maximum amount of blood drawn in a 24 hour period.
4. Patient or legal guardian must be able to speak and read at a 6th grade reading level.
5. Both male and female patients will be eligible
6. All races and ethnic backgrounds will be included
7. Relationships to proband: All patients with morphea will be included. A patient's family history will be reviewed and if there is a family history of morphea or systemic sclerosis then we will give the study patient the investigator's contact information and ask the family member to call the study team to answer any questions and enroll them in the study if they choose to do so.
8. Ability to give informed consent: Patients must be able to give informed consent or they will give assent with parent or guardian consent as a minor to be a part of the morphea registry.

Exclusion Criteria:

- Patients who have been coded as morphea (701.0), but do not have morphea/localized scleroderma (examples: steroid atrophy, acquired keratoderma, keloids, nephrogenic fibrosing dermopathy, systemic sclerosis, lichen sclerosis)

Max Age: 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Recruitment from clinic visits as well as from regional and national referrals.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2007-05 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Activity/damage measurement in morphea as scored on the Localized Scleroderma Cutaneous Assessment Tool (LoSCAT) | 5 years

SECONDARY OUTCOMES:
Quality of life scores measured by the Dermatology Life Quality Index (DLQI) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Jacobe, MD, MSCS, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center - Department of Dermatology, Dallas, Texas, United States

REFERENCES:
- See also: UTSW Morphea Registry Homepage — http://www.utsouthwestern.edu/education/medical-school/departments/dermatology/research/morphea-registry/index.html